CLINICAL TRIAL: NCT01776008
Title: A Phase II Trial of Neoadjuvant MK-2206 in Combination With Either Anastrozole if Postmenopausal or Anastrozole and Goserelin if Premenopausal in Women With Clinical Stage 2 or 3 PIK3CA Mutant Estrogen Receptor Positive and HER2 Negative Invasive Breast Cancer
Brief Title: Akt Inhibitor MK-2206 and Anastrozole With or Without Goserelin Acetate in Treating Patients With Stage II-III Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study did not pass Stage 1 interim analysis.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00080; NCI-2013-00080 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1139; MC1139 (Other: Mayo Clinic Cancer Center P2C); 9170 (Other: CTEP); N01CM00071 (NIH); N01CM00099 (NIH); P30CA015083 (NIH)
Record Dates: First submitted 2013-01-23; First posted 2013-01-25 (Estimated); Results first posted 2018-05-08 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Estrogen Receptor Positive; HER2/Neu Negative; Recurrent Breast Carcinoma; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — MK 2206; Anastrozole; Goserelin; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (MK2206, anastrozole, goserelin acetate) (Experimental): Patients receive Akt inhibitor MK-2206 PO on days 2, 9, 16, and 23; anastrozole PO daily on days 1-28; and goserelin acetate SC on day 1 (premenopausal patients only). Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt Inhibitor MK2206; Drug: Anastrozole; Drug: Goserelin Acetate; Other: Laboratory Biomarker Analysis; Procedure: Neoadjuvant Therapy; Other: Pharmacological Study; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Akt Inhibitor MK2206 — Given PO
  Other Names: MK2206
Drug: Anastrozole — Given PO
  Other Names: Anastrazole; Arimidex; ICI D1033; ICI-D1033; ZD-1033
Drug: Goserelin Acetate — Given SC
  Other Names: ZDX; Zoladex
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Neoadjuvant Therapy — Given before standard-care surgery
  Other Names: Induction Therapy; Neoadjuvant; Preoperative Therapy
Other: Pharmacological Study — Correlative studies
Procedure: Therapeutic Conventional Surgery — Undergo standard-care surgery

SUMMARY:
This phase II trial studies how well Akt inhibitor MK-2206 (MK-2206) and anastrozole with or without goserelin acetate works in treating patients with stage II-III breast cancer. MK-2206 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Estrogen can cause the growth of breast cancer cells. Hormone therapy using anastrozole and goserelin acetate may fight breast cancer by blocking the use of estrogen by the tumor cells. Giving MK-2206, anastrozole, and goserelin acetate together may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the pathologic complete response (pCR) rate of neoadjuvant MK-2206 (Akt inhibitor MK-2206) in combination with anastrozole (goserelin [goserelin acetate] is added if premenopausal) in women with clinical stage II or III phosphatidlinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha (PIK3CA) mutated estrogen receptor (ER)+/human epidermal growth factor receptor 2 (HER2)- breast cancer.

SECONDARY OBJECTIVES:

I. To determine the safety profile of neoadjuvant MK-2206 in combination with anastrozole (goserelin is added if premenopausal) in women with clinical stage II or III PIK3CA mutated ER+/HER2- breast cancer.

II. To estimate the rate of clinical response and radiologic response using the World Health Organization (WHO) criteria.

TERTIARY OBJECTIVES:

I. For pre and post-menopausal women separately, to examine serum estradiol levels prior to pre-registration, prior to registration, after 2 cycles of anastrozole plus MK-2206 (cycle 3 day 1) and pre surgery.

II. To examine the percent change in the apoptotic index after 2 weeks of combination therapy with MK-2206 and anastrozole (cycle 1 day 17) relative to apoptotic index after 4 weeks of treatment with anastrozole alone (pre MK-2206).

III. To examine the change in Ki67 levels after 2 weeks of combination therapy with MK-2206 and anastrozole (cycle 1 day 17) relative to that after 4 weeks of treatment with anastrozole alone (pre MK-2206).

IV. To estimate the proportion of patients whose Ki67 values is at most 10% after 2 weeks of combination therapy with MK-2206 and anastrozole (cycle 1 day 17) among those whose Ki67 was more than 10% or more after 4 weeks of treatment with anastrozole alone (pre MK-2206).

V. To examine the pharmacodynamic effect of MK-2206 in combination with anastrozole (or anastrozole in combination with goserelin) on PI3K pathway signaling using serially collected tumor specimens.

VI. To explore molecular mechanisms which could affect tumor response to combination MK-2206 and anastrozole (or anastrozole in combination with goserelin) in PIK3CA mutant ER+ breast cancer.

VII. To examine the PIK3CA mutation status in circulating plasma deoxyribonucleic acid (DNA) prior to and following therapy on serially collected peripheral blood (pre anastrozole, pre MK-2206, cycle 1 day 17, and at the time of surgery) and to correlate with tumor tissue PIK3CA status.

VIII. To examine PIK3CA mutation status of the residual cancer collected at the time of surgery post 4 cycles of neoadjuvant MK-2206 and anastrozole.

OUTLINE:

Patients receive Akt inhibitor MK-2206 orally (PO) on days 2, 9, 16, and 23; anastrozole PO daily on days 1-28; and goserelin acetate subcutaneously (SC) on day 1 (premenopausal patients only). Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Standard of care surgery (breast and axillary lymph node surgery) is performed 1-3 weeks following the last dose of Akt inhibitor MK-2206.

After completion of study treatment, patients are followed up for 30-60 days.

ELIGIBILITY:
Inclusion Criteria:

* Clinical T2-T4c, any N, M0 invasive ER+ (Allred score of 6-8) and HER2 negative (0 or 1+ by immunohistochemistry [IHC] or fluorescence in situ hybridization [FISH] negative for amplification) breast cancer, by American Joint Committee on Cancer (AJCC) 7th edition clinical staging, with the goal being surgery to completely excise the tumor in the breast and the lymph node;

  * Note: if the patient has invasive or ductal carcinoma in situ (DCIS) in the contralateral breast the patient is not eligible for this study
* >= 1 measurable lesion that is palpable, its size can be measured by bi-dimensional tape, ruler or caliper technique, and the minimum size of the largest tumor diameter is greater than 2.0 cm by imaging or physical examination
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Life expectancy > 4 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN
* Creatinine =< ULN OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine above institutional normal
* Patient with diabetes mellitus: fasting glucose =< 120 mg/dL and hemoglobin A1c (HbA1c) =< 8%
* Negative serum pregnancy test =< 7 days prior to pre-registration for women of childbearing potential
* Ability to understand and the willingness to sign a written informed consent document
* Patient is postmenopausal or premenopausal

  * NOTE: postmenopausal women, verified by

    * Bilateral surgical oophorectomy, or
    * No spontaneous menses >= 1 year or
    * No menses for < 1 year with follicle stimulating hormone (FSH) and estradiol levels in postmenopausal range, according to institutional standards or
  * Premenopausal women, verified by:

    * Regular menses or
    * FSH and estradiol levels in premenopausal range, according to institutional standards
* Willingness to provide biologic samples for PIK3CA sequencing and correlative studies
* Positive for PIK3CA mutation based on central laboratory testing
* In premenopausal women, serum estradiol level in postmenopausal range =< 7 days prior to registration

Exclusion Criteria:

* Any of the following for treatment of this cancer including:

  * Surgery
  * Radiation therapy
  * Chemotherapy
  * Biotherapy
  * Hormonal therapy
  * Investigational agent prior to study entry
* Receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-2206 or other agents used in this study
* Prior axillary lymph node sampling (sentinel lymph node biopsy or axillary lymph node dissection); NOTE: fine needle aspiration (FNA) of axillary lymph node is acceptable
* Invasive cancer or DCIS in the contralateral breast
* Receiving any medications or substances that are strong inhibitors or inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP450 3A4);

  * NOTE: oxidative metabolism of MK-2206 in human liver microsomes is catalyzed primarily by CYP3A4, although direct glucuronidation also occurs; at least 7 days washout period is required in patients who were previously taking strong inhibitors or inducers of CYP.450 3A4; patients who are currently taking moderate inhibitors or inducers of CYP450 3A4 are encouraged to switch to other medications that do not interact with CYP450 3A4
* Corrected QT interval (QTc) prolongation (defined as a QTc interval > 480 msec) or other significant electrocardiogram (ECG) abnormalities
* Receiving any medications or substances with risk of torsades de pointes; Note: medications or substances on the list "Drugs with Risk of Torsades de Pointes" are prohibited; medications or substances on the list "Drugs with Possible or Conditional Risk of Torsades de Pointes" may be used while on study with extreme caution and careful monitoring
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Uncontrolled symptomatic cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Any of the following:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential who are unwilling to employ adequate contraception
  * NOTE: breastfeeding should be discontinued if the mother is treated with MK-2206; women of childbearing potential must use two forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy; NOTE: HIV-positive patients on combination antiretroviral therapy are ineligible; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy
* Evidence of inflammatory cancer (clinical presentation of skin erythema involving more than one third of the breast or pathological evidence of dermal lymphatic involvement)
* Patients with known metastatic disease are excluded
* Current use of therapeutic anticoagulation therapy
* Previous excisional biopsy of the breast cancer
* Any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous [IV] alimentation, prior surgical procedures affecting absorption) that impairs patients ability to swallow MK-2206 tablets

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Ma, Principal Investigator — Mayo Clinic Cancer Center P2C
Locations (8):
- United States (8):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (MK2206, Anastrozole, Goserelin Acetate): Patients receive 150 mg Akt inhibitor MK-2206 PO on days 2, 9, 16, and 23; 1 mg anastrozole PO daily on days 1-28; and 3.6 mg goserelin acetate SC on day 1 (premenopausal patients only). Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (MK2206, Anastrozole, Goserelin Acetate)
Started | 16
Completed | 14
Not Completed | 2
Not completed — ineligible | 2

BASELINE CHARACTERISTICS:
Population: All patients registering were included in baseline description.
Arm/Group | Treatment (MK2206, Anastrozole, Goserelin Acetate)
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 57.5 [40 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response Rate
Description: Any woman whose Ki67 value ≤10% on cycle 1 day 17 of combination treatment who does not receive alternative treatment prior to surgery and has no histologic evidence of invasive tumor cells in the surgical breast specimen and the axillary lymph nodes is considered to have a pathological complete response (pCR). A ninety percent confidence interval for the true pathologic complete response rate will be calculated using the Duffy-Santer approach.
Time Frame: At time of surgery (up to 3 weeks after 4, 28-day cycles)
Population: All patients beginning protocol therapy and evaluable for primary endpoint were included in this analysis.
Measure: Number; unit: participants
Arm/Group | Treatment (MK2206, Anastrozole, Goserelin Acetate)
Number analyzed (Participants) | 16
participants | 0

2. Secondary Outcome: Clinical Response Rate
Description: The Clinical response rate is estimated by the number of patients whose disease meets the WHO criteria of complete or partial response based on physical examination divided by the total number of eligible patients. Complete Response (CR) is defined as the disappearance of all known disease based on measurements taken at the completion of neo-adjuvant therapy. Partial Response (PR) is defined as a 50% or greater decrease in the product of the bi-dimensional measurements of the lesion (total tumor size) between the pre-treatment measurements and the measurements taken at the completion of neo-adjuvant therapy. A ninety percent confidence interval for the true clinical response rate will be calculated using the Duffy-Santer approach.
Time Frame: Baseline to end of Cycle 4 (28 day cycles)
Population: Due to missing bi-dimensional measurements, clinical response could not be determined.
Arm/Group | Treatment (MK2206, Anastrozole, Goserelin Acetate)
Number analyzed (Participants) | 0

3. Secondary Outcome: Incidence of Adverse Events, Based on the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. For this endpoint, we are reporting the number of patients that reported a grade 3 or higher graded adverse event during neoadjuvent treatment. A complete list of all reported adverse events is in the Adverse Events section of the report.
Time Frame: Baseline to end of Cycle 4 (28 day cycles)
Population: All patients that registered and began neoadjuvant treatment were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (MK2206, Anastrozole, Goserelin Acetate)
Number analyzed (Participants) | 16
Participants
  Grade 3+ Adverse Event | 6
  Grade 4+ Adverse Event | 2

4. Secondary Outcome: Radiological Response Rate
Description: The Clinical response rate is estimated by the number of patients whose disease meets the WHO criteria of complete or partial response based on radiographic evaluation (mammogram or ultrasound) divided by the total number of eligible patients. Complete Response (CR) is defined as the disappearance of all known disease based on measurements taken at the completion of neo-adjuvant therapy. Partial Response (PR) is defined as a 50% or greater decrease in the product of the bi-dimensional measurements of the lesion (total tumor size) between the pre-treatment measurements and the measurements taken at the completion of neo-adjuvant therapy. A ninety percent confidence interval for the true clinical response rate will be calculated using the Duffy-Santer approach.
Time Frame: Baseline and completion of cycle 4 (28 day cycles)
Population: Due to missing pre-surgical scans, this endpoint could not be evaluated.
Arm/Group | Treatment (MK2206, Anastrozole, Goserelin Acetate)
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Change in Ki67 Levels
Time Frame: From 2 weeks of combination therapy with Akt inhibitor MK2206 and anastrozole (day 17 of course 1) to after 4 weeks of treatment with anastrozole alone
Population: Data was not collected
Arm/Group | Treatment (MK2206, Anastrozole, Goserelin Acetate)
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Percent Change in the Apoptotic Index
Time Frame: as for outcome 5
Population: Data was not collected.
Arm/Group | Treatment (MK2206, Anastrozole, Goserelin Acetate)
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Proportion of Patients Whose Ki67 Values is at Most 10%
Description: A 95% binomial confidence intervals will be constructed for the true proportion of patients whose pre Akt inhibitor MK2206 ki67 value is at most 10% as well as for the true proportion of patients with a C1D17 Ki67 value that is at most 10% among those patients whose pre Akt inhibitor MK2206 Ki67 was more than 10%.
Time Frame: as for outcome 5
Population: Data was not collected.
Arm/Group | Treatment (MK2206, Anastrozole, Goserelin Acetate)
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Serum Estradiol Levels
Time Frame: At baseline, following 4 weeks of anastrozole alone, day 1 of course 3, and at pre-surgery
Population: Data was not collected.
Arm/Group | Treatment (MK2206, Anastrozole, Goserelin Acetate)
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: The Pharmacodynamic Effect of Akt Inhibitor MK2206 in Combination With Anastrozole on the PI3K Pathway Activities, Assessed by Phosphoroproteomics and Immunohistochemistry Analysis on Serial Tumor Biopsies
Time Frame: Up to 3 weeks following the last dose of Akt inhibitor MK-2206
Population: Data was not collected.
Arm/Group | Treatment (MK2206, Anastrozole, Goserelin Acetate)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected after every cycle of treatment (28 day cycles) and up to 60 days after surgery.
Description: Adverse Events were collected after every cycle of treatment (28 day cycles) and up to 60 days after surgery.
Arm/Group | Treatment (MK2206, Anastrozole, Goserelin Acetate)
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (MK2206, Anastrozole, Goserelin Acetate) (N=16)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (MK2206, Anastrozole, Goserelin Acetate) (N=16)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (3)
Dry mouth (Gastrointestinal disorders) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 6 (9)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 14 (42)
Fever (General disorders) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (9)
Hyperglycemia (Metabolism and nutrition disorders) | 12 (34)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (3)
Headache (Nervous system disorders) | 2 (5)
Agitation (Psychiatric disorders) | 1 (3)
Libido decreased (Psychiatric disorders) | 1 (2)
Libido increased (Psychiatric disorders) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 1 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (20)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (15)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 (25)
Hot flashes (Vascular disorders) | 2 (4)
Hypertension (Vascular disorders) | 1 (2)
Vascular disorders - Other, specify (Vascular disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less